CLINICAL TRIAL: NCT01112306
Title: Long-term Single-arm Open-label Study, to Assess the Safety and Tolerability of ACT-293987 in Patients With Pulmonary Arterial Hypertension
Brief Title: ACT-293987 in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-065A303; 2009-014992-31 (EudraCT Number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-28 (Estimated); Results first posted 2022-09-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Open-label; PAH; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): ACT-293987, twice daily
  Interventions: Drug: ACT-293987

INTERVENTIONS:
Drug: ACT-293987 — Tablets, twice daily

SUMMARY:
Long-term, single-arm, multicenter, open-label extension, Phase 3 study, to evaluate the safety and tolerability of ACT-293987 in patients with PAH who participated in the double-blind study AC-065A302 (GRIPHON)

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated to the double-blind study AC-065A302 and either had a morbidity event or had completed the study as scheduled per protocol.
* Signed informed consent.

Exclusion Criteria:

* Patients who have started receiving prostacyclin (epoprostenol) or prostacyclin analogs (i.e., treprostinil, iloprost, beraprost) since the last study drug intake in AC-065A302/GRIPHON.
* Severe hepatic impairment (Child-Pugh C).
* Females who are pregnant or who plan to become pregnant during the study, or are breastfeeding.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results, such as drug or alcohol dependence, or psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2010-07-07 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Frey, Study Director — Actelion
Locations (157):
- United States (45):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Sacramento, California
  - Torrance, California
  - Newark, Delaware
  - Atlanta, Georgia
  - Augusta, Georgia
  - Austell, Georgia
  - Carmel, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Newark, New Jersey
  - Islandia, New York
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Bend, Oregon
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - York, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Corrientes
  - Córdoba
- Australia (10):
  - Adelaide
  - Bedford Park
  - Chermside
  - Concord
  - Darlinghurst
  - Fitzroy
  - Hobart
  - Murdoch
  - New Lambton
  - Parkville
- Austria (2):
  - Graz
  - Vienna
- Minsk, Belarus
- Belgium (2):
  - Brussels
  - Leuven
- Canada (8):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Santiago, Chile
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai
- Bogotá, Colombia
- Prague, Czechia
- Denmark (2):
  - Aarhus
  - Copenhagen
- France (4):
  - Bron
  - Le Kremlin-Bicêtre
  - Lille
  - Toulouse
- Germany (10):
  - Berlin
  - Cologne
  - Dresden
  - Giessen
  - Greifswald
  - Hanover
  - Heidelberg
  - Leipzig
  - Löwenstein
  - Regensburg
- Greece (3):
  - Alexandroupoli
  - Athens
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- India (3):
  - Ahmedabad
  - Chennai
  - Hyderabad
- Dublin, Ireland
- Israel (6):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Kuala Lumpur, Malaysia
- Mexico City, Mexico
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Rotterdam
- Lima, Peru
- Poland (4):
  - Gdansk
  - Krakow
  - Lodz
  - Otwock
- Romania (2):
  - Bucharest
  - Iași
- Russia (7):
  - Barnaul
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tomsk
  - Yekaterinburg
- Belgrade, Serbia
- Singapore, Singapore
- Slovakia (2):
  - Bratislava
  - Košice
- South Korea (2):
  - Incheon
  - Seoul
- Spain (2):
  - Barcelona
  - Madrid
- Sweden (4):
  - Gothenburg
  - Linköping
  - Umeå
  - Uppsala
- Switzerland (4):
  - Basel
  - Bern
  - Geneva
  - Lausanne
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Khon Kaen, Thailand
- Turkey (Türkiye) (3):
  - Adana
  - Istanbul
  - Izmir
- Ukraine (4):
  - Dnipro
  - Kharkiv
  - Kyiv
  - Lviv
- United Kingdom (2):
  - Glasgow
  - London

REFERENCES:
- [Derived] Galie N, Gaine S, Channick R, Coghlan JG, Hoeper MM, Lang IM, McLaughlin VV, Lassen C, Rubin LJ, Hsu Schmitz SF, Sitbon O, Tapson VF, Chin KM. Long-Term Survival, Safety and Tolerability with Selexipag in Patients with Pulmonary Arterial Hypertension: Results from GRIPHON and its Open-Label Extension. Adv Ther. 2022 Jan;39(1):796-810. doi: 10.1007/s12325-021-01898-1. Epub 2021 Oct 30. PMID 34727317

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Survival analysis was planned in subset of participants who received selexipag in main study (NCT01106014) and either entered or did not enter this open label (OL) study. Safety analysis including all-cause mortality was planned for OL safety set. Hence, all-cause mortality data is based on participants who received study drug (selexipag or placebo) in main study and entered this OL study. Participants who did not enter this OL study were not analyzed for all-cause mortality.
Groups:
- Selexipag: Participants with pulmonary arterial hypertension (PAH) who completed the double-blind AC-065A302 GRIPHON study (NCT01106014) or experienced a morbidity event in that study, entered in this open label (OL) study. Participants who received selexipag in GRIPHON continued to receive selexipag at the same dose (200 micrograms [mcg], twice daily [bid] up to 1600 mcg bid based on individual maximum tolerated dose) in this OL study. Participants who were on placebo or experienced a morbidity event in GRIPHON entered the titration period of this OL-study and received lowest dose of selexipag (200 mcg, bid) and dose was titrated up to 1600 mcg bid, based on the individual maximum tolerated dose. Each participant received study drug from Day 1 until the earliest of a) selexipag became commercially available in this indication in participant's country, b) sponsor decided to stop current study, or c) participant/investigator decided to discontinue study intervention (up to 10.5 years).
Period: Overall Study
Arm/Group | Selexipag
Started | 709
Completed | 424
Not Completed | 285
Not completed — Death | 175
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 31
Not completed — Other | 70

BASELINE CHARACTERISTICS:
Arm/Group | Selexipag
Number analyzed (Participants) | 709
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 590
  Male | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 171
  BLACK OR AFRICAN AMERICAN | 15
  HISPANIC | 87
  OTHER | 8
  WHITE | 428
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 20
  AUSTRALIA | 37
  AUSTRIA | 3
  BELARUS | 34
  BELGIUM | 17
  CANADA | 13
  CHILE | 31
  CHINA | 113
  COLOMBIA | 3
  CZECH REPUBLIC | 11
  DENMARK | 4
  FRANCE | 21
  GERMANY | 35
  GREECE | 6
  HUNGARY | 10
  INDIA | 15
  IRELAND | 4
  ISRAEL | 11
  ITALY | 4
  MALAYSIA | 2
  MEXICO | 20
  NETHERLANDS | 4
  PERU | 6
  POLAND | 7
  ROMANIA | 9
  RUSSIAN FEDERATION | 72
  SERBIA | 10
  SINGAPORE | 8
  SLOVAKIA | 1
  SOUTH KOREA | 11
  SPAIN | 8
  SWEDEN | 10
  SWITZERLAND | 2
  TAIWAN | 11
  THAILAND | 4
  TURKEY | 8
  UKRAINE | 35
  UNITED KINGDOM | 9
  UNITED STATES | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) up to 3 Days After Study Intervention Discontinuation
Description: An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. A TEAE is any AE temporally associated with the use of study drug (from study drug initiation until 3 days after study drug discontinuation), whether or not considered related to the study drug.
Time Frame: Up to 3 days after study drug discontinuation (Up to 10.5 years)
Population: The open label (OL) safety analysis set included all randomized participants who received at least 1 dose of selexipag or placebo in main GRIPHON study (AC-065A302; NCT01106014) and entered to this current GRIPHON OL study (AC-065A303; NCT01112306). Participants who did not enter GRIPHON OL were not in the scope of the OL safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 709
Participants | 684

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) up to 3 Days After Study Intervention Discontinuation
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Those SAEs occurring during study drug administration, that is, between study drug initiation and three days after study drug discontinuation, are defined as treatment-emergent SAEs.
Time Frame: Up to 3 days after study drug discontinuation (Up to 10.5 years)
Population: The OL safety analysis set included all randomized participants who received at least 1 dose of selexipag or placebo in main GRIPHON study (AC-065A302; NCT01106014) and entered to this current GRIPHON OL study (AC-065A303; NCT01112306). Participants who did not enter GRIPHON OL were not in the scope of the OL safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 709
Participants | 420

3. Primary Outcome: Number of Participants With TEAEs Leading to Permanent Discontinuation of Study Intervention
Description: as for outcome 1
Time Frame: Up to 10.5 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 709
Participants | 129

4. Secondary Outcome: Percentage of Alive Participants
Description: Percentage of alive participants were analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Baseline (Day 1), Months 3, 6, 9, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120
Population: Selexipag-treated set (STS): all participants who received at least 1 dose of selexipag in either main study (NCT01106014) or this OL study (NCT01112306). Survival analysis was planned in a subset of STS participants who received selexipag in main study, entered or did not enter this OL study. Here, "n" (number analyzed): participants at risk (alive and on study), analyzed at each specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selexipag
Number analyzed (Participants) | 574
Percentage of participants
  KM estimate at Baseline (Day 1) | 100 [100 to 100]
  KM estimate at Month 3: number analyzed (Participants) | 558
  KM estimate at Month 3 | 98.4 [97.0 to 99.2]
  KM estimate at Month 6: number analyzed (Participants) | 543
  KM estimate at Month 6 | 96.3 [94.4 to 97.6]
  KM estimate at Month 9: number analyzed (Participants) | 527
  KM estimate at Month 9 | 94.0 [91.7 to 95.7]
  KM estimate at Month 12: number analyzed (Participants) | 501
  KM estimate at Month 12 | 92.0 [89.4 to 94.0]
  KM estimate at Month 24: number analyzed (Participants) | 397
  KM estimate at Month 24 | 85.3 [82.0 to 88.0]
  KM estimate at Month 36: number analyzed (Participants) | 305
  KM estimate at Month 36 | 79.3 [75.4 to 82.6]
  KM estimate at Month 48: number analyzed (Participants) | 235
  KM estimate at Month 48 | 75.2 [70.9 to 78.9]
  KM estimate at Month 60: number analyzed (Participants) | 177
  KM estimate at Month 60 | 71.2 [66.5 to 75.3]
  KM estimate at Month 72: number analyzed (Participants) | 139
  KM estimate at Month 72 | 66.8 [61.6 to 71.4]
  KM estimate at Month 84: number analyzed (Participants) | 119
  KM estimate at Month 84 | 63.3 [57.8 to 68.3]
  KM estimate at Month 96: number analyzed (Participants) | 89
  KM estimate at Month 96 | 60.3 [54.4 to 65.7]
  KM estimate at Month 108: number analyzed (Participants) | 44
  KM estimate at Month 108 | 56.9 [50.3 to 62.9]
  KM estimate at Month 120: number analyzed (Participants) | 10
  KM estimate at Month 120 | 56.9 [50.3 to 62.9]

ADVERSE EVENTS:
Time Frame: Up to 10.5 years
Description: The open label (OL) safety analysis set included all randomized participants who received at least 1 dose of selexipag or placebo in main GRIPHON study (AC-065A302; NCT01106014) and entered to this current GRIPHON OL study (AC-065A303; NCT01112306). Participants who did not enter GRIPHON OL were not in the scope of the OL safety analysis set.
Arm/Group | Selexipag
All-Cause Mortality (participants affected / at risk) | 186/709
Serious Adverse Events (participants affected / at risk) | 420/709
Other Adverse Events (participants affected / at risk) | 598/709
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=709)
Anaemia (Blood and lymphatic system disorders) | 9
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 1
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2
Bone Marrow Failure (Blood and lymphatic system disorders) | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 2
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1
Pseudolymphoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 4
Acute Right Ventricular Failure (Cardiac disorders) | 11
Angina Pectoris (Cardiac disorders) | 1
Aortic Valve Stenosis (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 17
Atrial Flutter (Cardiac disorders) | 8
Atrial Tachycardia (Cardiac disorders) | 2
Atrioventricular Block (Cardiac disorders) | 1
Atrioventricular Block Complete (Cardiac disorders) | 3
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 13
Cardiac Failure (Cardiac disorders) | 8
Cardiac Failure Acute (Cardiac disorders) | 2
Cardiac Failure Chronic (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 4
Cardio-Respiratory Arrest (Cardiac disorders) | 5
Cardiogenic Shock (Cardiac disorders) | 9
Cardiopulmonary Failure (Cardiac disorders) | 8
Cardiorenal Syndrome (Cardiac disorders) | 1
Cardiovascular Insufficiency (Cardiac disorders) | 2
Chronic Left Ventricular Failure (Cardiac disorders) | 1
Chronic Right Ventricular Failure (Cardiac disorders) | 2
Cor Pulmonale (Cardiac disorders) | 2
Cor Pulmonale Acute (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 2
Left Ventricular Failure (Cardiac disorders) | 4
Myocardial Infarction (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Right Ventricular Dysfunction (Cardiac disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 93
Supraventricular Tachycardia (Cardiac disorders) | 4
Tricuspid Valve Incompetence (Cardiac disorders) | 1
Ventricular Tachyarrhythmia (Cardiac disorders) | 2
Dermoid Cyst (Congenital, familial and genetic disorders) | 1
Haemorrhagic Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1
Basedow's Disease (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Thyroiditis Subacute (Endocrine disorders) | 1
Astigmatism (Eye disorders) | 1
Diabetic Retinopathy (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal Hernia (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 6
Chronic Gastritis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 12
Diverticular Perforation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 9
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus Paralytic (Gastrointestinal disorders) | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 1
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Obstructive Pancreatitis (Gastrointestinal disorders) | 1
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Catheter Site Erythema (General disorders) | 1
Catheter Site Thrombosis (General disorders) | 1
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 7
Death (General disorders) | 3
Drowning (General disorders) | 1
Drug Ineffective (General disorders) | 1
Drug Interaction (General disorders) | 1
Euthanasia (General disorders) | 1
Fatigue (General disorders) | 1
Gait Disturbance (General disorders) | 1
Generalised Oedema (General disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 8
Oedema Peripheral (General disorders) | 4
Organ Failure (General disorders) | 1
Peripheral Swelling (General disorders) | 1
Pyrexia (General disorders) | 5
Sudden Cardiac Death (General disorders) | 3
Sudden Death (General disorders) | 14
Systemic Inflammatory Response Syndrome (General disorders) | 1
Withdrawal Syndrome (General disorders) | 1
Bile Duct Stone (Hepatobiliary disorders) | 1
Cardiac Cirrhosis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis Acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Amyloidosis (Immune system disorders) | 1
Abscess Bacterial (Infections and infestations) | 1
Abscess Limb (Infections and infestations) | 1
Actinomycotic Pulmonary Infection (Infections and infestations) | 1
Anal Abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Appendicitis Perforated (Infections and infestations) | 1
Atypical Pneumonia (Infections and infestations) | 1
Bacterial Abdominal Infection (Infections and infestations) | 1
Bacterial Sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 11
Cellulitis (Infections and infestations) | 6
Clostridium Difficile Colitis (Infections and infestations) | 1
Colonic Abscess (Infections and infestations) | 1
Complicated Appendicitis (Infections and infestations) | 1
Corona Virus Infection (Infections and infestations) | 4
Cystitis (Infections and infestations) | 1
Dengue Fever (Infections and infestations) | 1
Disseminated Tuberculosis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Enterobacter Sepsis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Escherichia Sepsis (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis Clostridial (Infections and infestations) | 1
Gastroenteritis Norovirus (Infections and infestations) | 1
Gastrointestinal Infection (Infections and infestations) | 1
H1n1 Influenza (Infections and infestations) | 1
Haematoma Infection (Infections and infestations) | 1
Haemorrhagic Pneumonia (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Infective Tenosynovitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 8
Lung Infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 2
Osteomyelitis (Infections and infestations) | 1
Otitis Media Bacterial (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 3
Peritonitis Bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 50
Pneumonia Bacterial (Infections and infestations) | 2
Pneumonia Viral (Infections and infestations) | 3
Postoperative Wound Infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 2
Pyoderma (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 10
Septic Shock (Infections and infestations) | 3
Sialoadenitis (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Staphylococcal Sepsis (Infections and infestations) | 2
Tracheobronchitis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 4
Viral Infection (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Accident (Injury, poisoning and procedural complications) | 1
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 3
Concussion (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 8
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2
Fractured Sacrum (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1
Poisoning (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1
Reactive Gastropathy (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 2
Skin Laceration (Injury, poisoning and procedural complications) | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 3
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Anticoagulation Drug Level above Therapeutic (Investigations) | 1
Biopsy Kidney (Investigations) | 1
Blood Uric Acid Increased (Investigations) | 1
Catheterisation Cardiac (Investigations) | 2
Haemoglobin Decreased (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 2
Investigation (Investigations) | 1
N-Terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 1
Precancerous Cells Present (Investigations) | 1
Prothrombin Time Prolonged (Investigations) | 1
Transplant Evaluation (Investigations) | 1
Weight Decreased (Investigations) | 1
Fluid Overload (Metabolism and nutrition disorders) | 3
Fluid Retention (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Fracture Malunion (Musculoskeletal and connective tissue disorders) | 1
Haematoma Muscle (Musculoskeletal and connective tissue disorders) | 1
Mixed Connective Tissue Disease (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Still's Disease (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoid Tumour of the Stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to the Mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nodal Marginal Zone B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Germ Cell Teratoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid Artery Occlusion (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Intracranial Haematoma (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 18
Transient Ischaemic Attack (Nervous system disorders) | 1
Vocal Cord Paralysis (Nervous system disorders) | 1
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5
Acute Psychosis (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Drug Dependence (Psychiatric disorders) | 1
Major Depression (Psychiatric disorders) | 2
Suicide Attempt (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 6
Chronic Kidney Disease (Renal and urinary disorders) | 3
Cystitis Haemorrhagic (Renal and urinary disorders) | 1
Glomerulonephritis Chronic (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Ischaemic Nephropathy (Renal and urinary disorders) | 1
Lupus Nephritis (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 4
Renal Haematoma (Renal and urinary disorders) | 1
Renal Impairment (Renal and urinary disorders) | 1
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Lower Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Lupus Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Alveolar Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 169
Pulmonary Artery Aneurysm (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Artery Dilatation (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2
Balloon Atrial Septostomy (Surgical and medical procedures) | 1
Benign Breast Lump Removal (Surgical and medical procedures) | 1
Breast Conserving Surgery (Surgical and medical procedures) | 1
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1
Coronary Angioplasty (Surgical and medical procedures) | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 1
Drug Therapy (Surgical and medical procedures) | 1
Fasciotomy (Surgical and medical procedures) | 1
Gastric Bypass (Surgical and medical procedures) | 1
Heart and Lung Transplant (Surgical and medical procedures) | 2
Hip Arthroplasty (Surgical and medical procedures) | 1
Knee Operation (Surgical and medical procedures) | 1
Lung Transplant (Surgical and medical procedures) | 5
Nephrectomy (Surgical and medical procedures) | 1
Ovarian Cystectomy (Surgical and medical procedures) | 1
Packed Red Blood Cell Transfusion (Surgical and medical procedures) | 1
Percutaneous Coronary Intervention (Surgical and medical procedures) | 1
Rehabilitation Therapy (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Varicose Vein Operation (Surgical and medical procedures) | 1
Vascular Operation (Surgical and medical procedures) | 1
Circulatory Collapse (Vascular disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 6
Hypovolaemic Shock (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
Superior Vena Cava Perforation (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selexipag (N=709)
Anaemia (Blood and lymphatic system disorders) | 65
Palpitations (Cardiac disorders) | 43
Diarrhoea (Gastrointestinal disorders) | 209
Nausea (Gastrointestinal disorders) | 135
Vomiting (Gastrointestinal disorders) | 74
Fatigue (General disorders) | 44
Oedema Peripheral (General disorders) | 90
Bronchitis (Infections and infestations) | 59
Nasopharyngitis (Infections and infestations) | 88
Upper Respiratory Tract Infection (Infections and infestations) | 84
Urinary Tract Infection (Infections and infestations) | 42
Hypokalaemia (Metabolism and nutrition disorders) | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 65
Myalgia (Musculoskeletal and connective tissue disorders) | 68
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 78
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 130
Dizziness (Nervous system disorders) | 71
Headache (Nervous system disorders) | 328
Cough (Respiratory, thoracic and mediastinal disorders) | 80
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 76
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 68
Flushing (Vascular disorders) | 49
Hypotension (Vascular disorders) | 38

LIMITATIONS AND CAVEATS:
The study had an open-label, uncontrolled design. Additional pulmonary arterial hypertension (PAH)-specific treatments were introduced in a limited percentage of participants and during a limited period of time. The study had a variable study duration across countries/territories depending on the availability of commercial selexipag. Limited safety data reporting was done in participants in China due to the human genetic resources (HGR) regulation finding after 20-December-2019.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01112306/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT01112306/SAP_001.pdf